CLINICAL TRIAL: NCT01731106
Title: Cerebral Autoregulation in Non Neurological Critical Patients.
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment rate
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Rafael Fernandez, Physician Doctor, Althaia Xarxa Assistencial Universitària de Manresa
Other Study IDs: Fundacio Unio CEIC 12/18
Record Dates: First submitted 2012-11-13; First posted 2012-11-21 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Critical Illness; Complication of Ventilation Therapy; Systemic Inflammatory Response Syndrome; Failed Moderate Sedation During Procedure, Sequela
MeSH Terms: conditions — Critical Illness; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for biomarkers at admision, 72 hours and 7 days.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Brief Summary Cerebral Autoregulation is a well known physiological response to blood pressure changes to maintain the cerebral perfusion. The critically ill patients are submitted to different situations that can impair the cerebral autoregulation as sepsis, sedation drugs and mechanical ventilation.

The delirium on ICU has been described as a bad prognosis factor, increasing the mortality and length of stay. The physiopathology of delirium has been related to cerebral perfusion. The delirium has been related to long term cognitive impairment.

Material and Methods:

This is a physiological prospective study that will be done in a 14 bed medical-surgical ICU. The investigators will enroll 100 ventilated patients, septic and non-septic. The investigators will measure cerebral autoregulation every 48-72 hours from admission on ICU. Neurological biomarkers (Neurological Specific Enolase, S100 beta and Vascular Endothelial Growing Factor) will be done at inclusion, 72 hours and 7 days. Clinical data, delirium presence, analytic data and ventilatory parameters will be registered every day.

At hospital discharge, a psychologist will do a cognitive evaluation using specific tests. The cognitive evaluation will be repeated at 3, 6 and 12 months.

Anticipate results:

Some items like mechanical ventilation, sepsis and sedation can impair cerebral autoregulation. The impairment of cerebral autoregulation is related to delirium in ICU and long cognitive impairment.

DETAILED DESCRIPTION:
Introduction:

Cerebral Autoregulation (CA) is the physiological strategy used for the brain to maintain the cerebral blood flow constant during blood pressure (BP) changes. The evaluation of CA dynamic and static models has been described in the literature. The coefficient Sx and the Mx are one of the validated dynamic methods. These coefficients are obtained from the correlation between BP and Middle Cerebral Artery (MCA) velocity measured using Transcranial Doppler (TCD). Correlation values higher than 0.3 reflect an impairment of CA.

The incidence of CA impairment in the Intensive Care Unit (ICU) is not well described. Neither, risk factors or clinical situations that precipitate CA impairment have been studied.

Mechanical Ventilation (MV) is a common treatment in the ICU. The main difference is the positive pressure administrated to the lungs instead of the negative pressure in spontaneous breathing. The positive pressure applied in the alveoli causes a local and systemic inflammatory response. Lung injuries are well described due to MV. Some studies relate changes in the Intracranial Pressure (ICP) and Cerebral Perfusion Pressure (CPP) with the Positive End- Expiratory Pressure in neurological patients. Also changes in the MCA velocity have been described with MV. The studies speculate that the changes are related to the intrathoracic positive pressure. However, all studies are in patients with acute neurological pathology.

In the ICU sedation drugs are often used to guarantee patient comfort in the MV. The BIS ® device is used for monitoring sedation level based on the electroencephalogram drawing. Recent studies analyse the influence of this drugs on CA in healthy volunteers. However, no studies have described the effects of long sedations like usually occurs in ICU.

The incidence of delirium in the ICU has been described as 50%. In mechanically ventilated patients the incidence increases to 80%. Delirium is considered an independent factor of bad prognosis. It increases the days under mechanical ventilation, hospital length of stay, the dependence at discharge and the risk of death. Because of that, it has a high impact in health and in economic cost. However it is an underdiagnosed illness due to the absence of ICU protocols for the correct diagnosis. The scale Confusion Assessment Method for ICU (CAM - ICU) is the validated tool for the screening and it is used by the nurses and physicians.

The long term cognitive impairment is well described in patients admitted in the ICU. A recent study followed-up the patients subjected to mechanical ventilator who had developed delirium. They use the Mini-mental State Examination Score and they found that at 3 month following-up 61% patients had severe cognitive impairment and 17% a moderate impairment. At 12 months the 36% of patients still had a severe impairment and the 35% a moderate impairment. The developing of delirium during the ICU admission is considered a risk factor for long term cognitive impairment.

Sepsis has been also related with cognitive impairment. Iwashyna et al, published that patients with basal moderate cognitive impairment who survived a severe infection, had higher probability of getting worse compared to patients who were admitted for other reasons.

Some biomarkers for neurological damage are well known. The S100B protein, present in the calcium canal of glial cells, and the Neurological Specific Enolase (NSE), an enzyme that participates in neurological glucolysis are increased in patients with Brain Trauma, cerebral ischemia or bleeding. In older patients with delirium the levels of S100B are also increased, but not the NSE levels. In critical patients the S100B and NSE have been used for delirium and cognitive impairment markers. However, the publications have been contradictories. Most of them find high levels of S100Bin septic and postoperative patients who developed delirium, but in some studies no significant differences have been seen. NSE has not relation with delirium in septic patients, however, after cardiac surgery with extracorporeal circulation both markers, S100B and NSE, are good predictors of delirium and cognitive impairment at 6 months.

Vascular Endothelial Growing Factor (VEGF) takes part in the vascular and cerebral regeneration in the neurological system. It is considered a neuronal protector. Cerebral hypoxia stimulates the expression of VEGF for starting the vascular neogenesis. No studies related VEGF with delirium in the critical patient. Assuming that hypoxia and ischemia can develop delirium in the ICU, the VEGF levels may be augmented.

Hypothesis:

The critical patient under mechanical ventilation can have impaired CA due to situation as sepsis and multiorgan failure. The CA impairment can be related to sedation, pressors or some co-morbidity.

Primary objective:

1. To determinate the CA impairment in critically ill patient.

Secondary objectives:

1. To describe evolving patterns of CA in the critically ill patient.
2. To describe the influence of MV, sedation and sepsis on CA.
3. To analyze the relation between CA impairment and delirium in the ICU and long term cognitive impairment.
4. To determinate the long term cognitive status of patients who had CA impairment during the ICU admission.
5. To determinate the levels and kinetic evolution, and prognosis power of the biomarkers S100B, NSE and VEGF in critically ill patients.
6. To describe the influence of CA impairment on mortality.

Material and methods:

Study Field This is a physiological observational prospective study done in a University Hospital of 400 beds approximately. The study will take place in a medical-surgical ICU of 14 beds.

Consecutive enrolment of patients admitted on Fundació Althaia ICU of Manresa, Spain.

Methods:

Cerebral autoregulation analysis The investigators will use TCD to determinate CA situation. A continuous monitoring of MCA velocity and simultaneous invasive arterial pressure will be done every 48-72 hours during admission and when the patient is under MV. The investigators will calculate the Mx and Sx coefficients, defined as Pearson correlation between the average of mean (Mx) and systolic (Sx) MCA velocity and average of the values of arterial pressure waveform every 3 minutes. The software used is DWL Compumedics Monitoring ® to measure MCA velocity and arterial pressure waveform every 1 millisecond. The monitoring test will take between 20 minutes and 1 hour time.

The sedation depth will be continuous monitored using Bispectral Index System (BIS) of Covidien ®. Ramsay scale will be registered every 6 hours by nurses.

Cognitive evaluation After the discharge from the hospital the cognitive situation will be evaluated using neuropsychological tests. A medical psychologist of Fundació Althaia Psychiatry Service will do the evaluation.

The test grouping has been designed following the recommendation for medical population. Two or more of these tests under 1.5 SD general population standards will be considered as cognitive impairment. The test used includes psychometric tools for neuropsychological evaluation:

* Attention and velocity of processing
* Selective attention: Trail Making Test Part A; direct numbers (WMS-III).
* Divide attention and velocity of processing: Trail Making Test Part B; Symbol test and numbers.
* Memory:
* Immediate verbal memory: direct numbers (WSM - III), learning: word list I (WMS- III).
* Short term verbal memory (WMS - III)
* Long term verbal memory (WMS - III)
* Short term visual memory (WMSD - III)
* Long term visual memory (WMS - III)
* Language:
* Verbal nomination for visual confrontation (Boston nomination test)
* Verbal comprehension (Token test)
* Visual-space and visual-construction function (WAIS - III)
* Executive function:
* Concept formation and cognitive flexibility (WSCT)
* Memory of work: inverse numbers (WMS - III)
* Verbal fluency.
* Previous performance estimation: vocabulary (WAIS - III). Depressive and psychotic evaluation While the long term cognitive impairment evaluation, Depressive symptomatology will also be evaluated using the Beck Inventory. The psychotic evaluation will be carried out using the Brief Psychiatric Evaluation Scale.

S100B, NSE and VEGF levels At inclusion time the levels of biomarkers S100B, NSE and VEGF will be determined. The investigators will repeat the samples at 72 hours and 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old of age.
* Patients under mechanical ventilation and/or sedation drugs and/or severe sepsis as defined on international criteria.
* Patients with arterial line.

Exclusion Criteria:

* Acute neurological pathology.
* Absence of arterial line.
* Severe haemodynamic instability defined as Mean Arterial Pressure (MAP) lower than 70 mmHg even with pressors.
* Absence of temporal bone window for doing TCD.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admited on the ICU that need mechanical ventialtion
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
To describe the incidence of impairment of cerebral autoregulation in critically ill patients. | 7 days

SECONDARY OUTCOMES:
To describe the incidence of delirium in critically ill patients with or without impairment of cerebral autoregulation | 30 days
To describe the long term cognitive impariment in critically ill patients. | 3, 6 and 12 months

OTHER OUTCOMES:
To describe the survival of patients who have impairment of cerebral autoregulation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez, Ph, MD, Study Director — Head of Department
Locations (1):
- Carles Subira Cuyas, Manresa, Barcelona, Spain